CLINICAL TRIAL: NCT02133313
Title: Icodextrin Effects on Glucose Transporter Activation and Mediators of Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Eric Wallace, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: ICO-X140206005
Record Dates: First submitted 2014-04-30; First posted 2014-05-08 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: End Stage Renal Disease
Keywords: Peritoneal Dialysis; Peritoneal Fibrosis; Glucose Transporters
MeSH Terms: conditions — Kidney Failure, Chronic; Peritoneal Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Biospecimens will be retained. Cells harvested from spent peritoneal dialysate will have RNA isolated and then cDNA will be preserved.
  Supernatent of spent peritoneal dialysate will be kept.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peritoneal Dialysis Patients: Patients on Peritoneal Dialysis

SUMMARY:
The time on peritoneal dialysis may be limited for a significant number of patients that use this modality of renal replacement therapy due to the inability of the peritoneal membrane to clear solutes or achieve adequate ultrafiltration, termed peritoneal membrane failure (PMF). This can be devastating for patients who have become accustomed to the quality of life provided by peritoneal dialysis and who otherwise have done well on this therapy. There is clinical evidence suggesting that icodextrin preserves the peritoneal membrane transport characteristics which may be linked to reduced cumulative glucose exposure of the peritoneal mesothelial cells. Theories to explain the role of dextrose in PMF have focused for the most part on the high intracellular concentrations of glucose without consideration to the potential pathogenic role of the glucose transporters which allow glucose entry into the cell. Experimental evidence in non-mesothelial cell lines indicate that some cellular processes that occur under high glucose conditions may not be related to intracellular glucose metabolism but to the type of glucose transporter allowing glucose entry. 3,4 However, little is known about these glucose transporters in peritoneal mesothelial cells and their potential role in the development of PMF.

We hypothesize the following

* The presence of Sodium Glucose Co-transporter (SGLT1) on peritoneal mesothelial cells plays a role in PMF under hyperglycemic conditions.
* Regulation of pro-fibrotic mediators such as reactive oxidative species,transforming growth factor β, and vascular endothelial growth factor are modulated by SGLT1 activation by glucose rather than glucose metabolism or concentration.
* Icodextrin does not activate the SGLT1 transporter establishing a mechanism that may explain the beneficial effects of icodextrin on peritoneal membrane transport.

DETAILED DESCRIPTION:
Participants enrolled in this study will have pertinent clinical information entered into a database. Participants will then have spent peritoneal dialysate collected at least every 6 months and analyzed for markers of fibrosis. Patients undergoing a special type of peritoneal dialysis start call urgent start peritoneal dialysis will have spent peritoneal dialysate collected more frequently at the start of peritoneal dialysis and then every 6 months. The results from the analysis of the peritoneal dialysate will then be correlated with data in the patient registry.

Quality assurance- As this is a single center trial all data will be monitored by the PI. Data will be entered in a prospective manner into the database by a research coordinator. Every 6 months data will be checked for accuracy by comparing to data collected for routine clinical purposes by both the home dialysis unit which tracks all hospitalizations, peritonitis, exit site infections, technique failures. As well as the dialysis access database maintained by the University of Alabama at Birmingham.

Source data verification- Data will come from both the history and physical of the primary investigator as well as electronic medical records at the University of Alabama at Birmingham and Falcon Electronic Health Record from Davita.

Data Dictionary is as follows. Variable / Field Name study_id Is the patient restarting Peritoneal dialysis after stopping If the patient is restarting are they restarting with the same catheter or a new catheter Date of 1st Access Length of time catheter placed prior to use How was the catheter placed: Surgically vs. Interventional Radiology Open versus laparoscopic Lysis of Adhesions Omentopexy Type of PD Catheter Has the patient had a second access procedure Medical Record Number Davita Medical Record Number Person Entering Data first_name last_name Date of Birth sex race address Is the patient new to dialysis? Has the patient previously been on peritoneal dialysis. transfer Why was peritoneal dialysis stopped. Type of Start: Urgent start versus traditional start Anuric Urgent Start: Inpatient or Outpatient Admit Date for PD Initiation Date of Discharge for pd initiation Did the patient require hemodialysis during urgent start period Indication for Hemodialysis Number of Hemodialysis sessions Nonsurgical catheter issues Date of PD start Age at PD start Date of PD graduation Length of time to PD graduation Reason for Urgent start PD first_dialysis_modality Predialysis education type_predialysis_education Glomerular filtration rate at time of PD start Has the patient stopped PD Did the patient stop Peritoneal dialysis or did they transfer out? Date PD was stopped Length of time on dialysis Age PD stopped Reason PD stopped When the patient transferred, did they transfer with an access or a permacath Cause of death Cause of End Stage Renal Disease (ESRD) Comorbidities Has the patient had a kidney transplant Previous abdominal surgeries? Type of previous abdominal surgeries height Indication for Peritoneal Equilibration Test (PET Date of PET Type of PET 2 hour D/P Creatinine 4 hour D/P Creatinine Transporter type 2 hour D/D0 Glucose 4 hour D/D0 Glucose Initial PET glucose PD Glucose 4 hours Glucose Absorption PET Drain Volume Ultrafiltration PD Sodium 0 Hour PD Sodium 1 Hour PD Sodium 2 hour PD Sodium 4 Hour Serum Sodium Minimum PD Sodium Level Systolic Blood Pressure Diastolic Blood Pressure Mean Arterial Pressure Weight Body Mass Index Hemoglobin Albumin Ferritin Iron Transferrin Saturation Hemoglobin A1c Creatinine Potassium BUN Sodium Hco3 Total Protein total cholesterol HDL LDL Vitamin D 25 Phosphorus Calcium PTH Kt/V Does the patient have a last fill Icodextrin versus dianeal Midday Total Liters per day Total Liters Total 6 month glucose exposure Is the patient on icodextrin Date of Icodextrin start Length of time on icodextrin Kt/v prior to icodextrin Kt/V after icodextrin Reason icodextrin stopped Date Icodextrin stopped Length of time on icodextrin Has the patient had peritonitis Date of infection Polymicrobial Pathogen Gram Positive Methicillin Resistant Gram Negative Ciprofloxacin Resistant Fungal Did the patient have antibiotics prior to fungal peritonitis What antibiotic Did the patient receive fungal prophylaxis Is this relapsing or recurrent Has the patient been hospitalized Date of admission Length of time to first admission Date of Discharge Length of stay Reason for admit Hospitalization Outcome Cause of death

Standard Operating Procedures: Patient recruitment will be from the University of Alabama at Birmingham Home Dialysis unit.

Sample size: As there are no data on which to base the power calculation for this unique study on glucose transporters and their role in peritoneal membrane fibrosis, descriptive statistics will be used to gain insight into the proposed research questions. Continuous variables will be summarized with mean and standard deviation or median and interquartile range depending on the distribution. Categorical variables will be summarized with frequency and percentage.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* On Peritoneal Dialysis

Exclusion Criteria:

* none

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over the age of 19 on Peritoneal Dialysis at the University of Alabama at Birmingham
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2014-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in glucose transporter expression on peritoneal mesothelial cells | baseline to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Wallace, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Home Dialysis Unit (Red Mountain Home Dialysis), Birmingham, Alabama, United States

REFERENCES:
- [Background] Davies SJ, Phillips L, Naish PF, Russell GI. Peritoneal glucose exposure and changes in membrane solute transport with time on peritoneal dialysis. J Am Soc Nephrol. 2001 May;12(5):1046-1051. doi: 10.1681/ASN.V1251046. PMID 11316864
- [Background] Davies SJ, Brown EA, Frandsen NE, Rodrigues AS, Rodriguez-Carmona A, Vychytil A, Macnamara E, Ekstrand A, Tranaeus A, Filho JC; EAPOS Group. Longitudinal membrane function in functionally anuric patients treated with APD: data from EAPOS on the effects of glucose and icodextrin prescription. Kidney Int. 2005 Apr;67(4):1609-15. doi: 10.1111/j.1523-1755.2005.00243.x. PMID 15780118
- [Background] Balteau M, Tajeddine N, de Meester C, Ginion A, Des Rosiers C, Brady NR, Sommereyns C, Horman S, Vanoverschelde JL, Gailly P, Hue L, Bertrand L, Beauloye C. NADPH oxidase activation by hyperglycaemia in cardiomyocytes is independent of glucose metabolism but requires SGLT1. Cardiovasc Res. 2011 Nov 1;92(2):237-46. doi: 10.1093/cvr/cvr230. Epub 2011 Aug 22. PMID 21859816
- [Background] Palazzo M, Gariboldi S, Zanobbio L, Selleri S, Dusio GF, Mauro V, Rossini A, Balsari A, Rumio C. Sodium-dependent glucose transporter-1 as a novel immunological player in the intestinal mucosa. J Immunol. 2008 Sep 1;181(5):3126-36. doi: 10.4049/jimmunol.181.5.3126. PMID 18713983
- [Background] Schroppel B, Fischereder M, Wiese P, Segerer S, Huber S, Kretzler M, Heiss P, Sitter T, Schlondorff D. Expression of glucose transporters in human peritoneal mesothelial cells. Kidney Int. 1998 May;53(5):1278-87. doi: 10.1046/j.1523-1755.1998.00899.x. PMID 9573543
- [Background] Fischereder M, Schroppel B, Wiese P, Fink M, Banas B, Schmidbauer S, Schlondorff D. Regulation of glucose transporters in human peritoneal mesothelial cells. J Nephrol. 2003 Jan-Feb;16(1):103-9. PMID 12649541